CLINICAL TRIAL: NCT02290444
Title: Effects of Adrenocorticotropic Hormone (ACTHAR Gel) on Recovery From Cognitive Relapses in Multiple Sclerosis
Brief Title: Effects of Acthar on Recovery From Cognitive Relapses in MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ralph H.B. Benedict, Professor of Neurology and Psychiatry, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 465028
Record Dates: First submitted 2014-10-23; First posted 2014-11-14 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: Acute Relapsing Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitively Relapsing Patients (Experimental): For individuals experiencing cognitive relapses/exacerbations, 5ml/80 IU of Adrenocorticotropic Hormone will be administered through either subcutaneous or intramuscular self-injection (selected by the patient) for 5-days.
  Interventions: Drug: Adrenocorticotropic Hormone
- Stable Multiple Sclerosis Patients (No Intervention): Individuals whose Multiple Sclerosis is currently in a stable state (not currently or recently exacerbating) are age-matched with relapsing MS patients. There is no intervention for individuals with MS whose are currently in a stable state.

INTERVENTIONS:
Drug: Adrenocorticotropic Hormone — Acthar Gel will be administered in accordance with the recommendations set forth in the package insert. The dosage may be individualized according to the medical condition of each patient. Frequency and dose of the drug may be determined by considering the severity of the disease and the initial response of the patient.
  Other Names: Acthar gel
  Arms: Cognitively Relapsing Patients

SUMMARY:
The purpose of this study is to evaluate the effect of a medication called Acthar on recovery from multiple sclerosis-related relapses that impact cognition.

DETAILED DESCRIPTION:
This is a prospective, open-label study of Acthar administered as treatment for an acute cognitive relapse. Primary and secondary endpoints will be collected prior to Acthar administration and at 3-month follow-up. Comparison will be made to a stable MS control group.

The objectives of the study are:

1. To replicate prior findings with steroid therapy for MS patients for cognitive relapses, using instead Acthar Gel as the treating agent. The investigators will determine if the decrease on cognitive endpoints at the time of relapse exceeds that of stable MS controls.
2. To compare the effects above to a previously acquired dataset of relapsing patients treated with steroids. This is a quasi-experimental design in so far as the steroid treated group data were previously acquired in a separate study.

The primary hypothesis of the study is that, due to the enhanced melanocortin response in Acthar the recovery from cognitive changes occurring during cognitively focused relapse will be significant compared to stable MS patients matched on age, time since testing, and cognitive performance on the SDMT.

Target enrollment for the Acthar treatment group will be 30 MS patients under care at the Jacobs Neurological Institute with existing neuropsychological baseline in the past four years in whom a cognitive relapse or new supratentorial GAD enhancing lesion(s) on MRI have been identified. Cognitive relapse will be identified based on clinical presentation of acute worsening of cognitive symptoms in the domains of processing speed, concentration, episodic memory, working memory, and/or fatigue. Patients whose clinical MRI indicate new active GAD enhancing lesions will be screened for the presence of self-perceived cognitive decline, without new physical symptoms. Thirty (30) clinically stable MS patients matched on age, time since testing, and cognitive performance on the SDMT will be recruited from the pool of patients with existing cognitive baselines.

ELIGIBILITY:
Inclusion Criteria:

1. Males/Females between 18 and 65 years of age who are capable of understanding and complying with the protocol (ie. have completed at least a 9th grade education and are fluent English).
2. Have a diagnosis of Relapsing Remitting MS (RRMS) or early Secondary Progressive MS (SPMS) as per revised McDonald's Criteria.
3. Have an Expanded Disability Severity Scale (EDSS) of ≤ 7.0.
4. Have had valid neuropsychological testing (NP) within the past 4 years
5. Experiencing an acute cognitive relapse identified by a clinical care provider as a.) a cognitive symptom of recent origin developing over 48 hours, or b.) supratentorial GAD enhancing lesions on MRI with confirmed cognitive decline.

   * Confirmation of cognitive decline will be obtained by administering the Symbol Digit Modalities Test (SDMT) as a screening procedure for the study and comparing it to scores obtained within 4 years (see inclusion criteria #4). Participants qualify if a raw point change on the SDMT greater than or equal to -3 points is detected.
6. Are capable of performing the requirements of neuropsychological (NP) testing, including near visual acuity 20/70 or better with correction.
7. Have given written informed consent prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care.

Exclusion Criteria:

1. Are found to have evidence on MRI of new lesions in the brainstem, spinal cord, or optic nerve.
2. Have clear new physical signs or symptoms that are referable to the cord, brainstem or optic nerve.
3. Have cognitive deficits/impairment caused by concomitant medication usage, or are attributable to another medical condition or significant neurological/psychological disease.
4. Have evidence of current major depression as determined by a positive Beck Depression Inventory-Fast Screen (BDI-FS) and clinician interview.
5. Patients with changes to medications known to influence cognition (narcotics, stimulants, etc.) or disease modifying therapy within one month of study initiation (or within a time frame deemed high risk by treating physician) will be excluded.
6. Are taking any medication, or have any medical condition contraindicated with Acthar.
7. Presence of current infections as determined by clinician interview.
8. Are currently nursing, intentionally seeking pregnancy, or deemed at-risk for unplanned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-08; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph HB Benedict, PhD, Principal Investigator — University of Buffalo-State University of New York
Locations (1):
- University at Buffalo-State University of New York, Department of Neurology, Buffalo General Hospital, Buffalo, New York, United States

REFERENCES:
- [Background] Benedict RH, Zivadinov R. Predicting neuropsychological abnormalities in multiple sclerosis. J Neurol Sci. 2006 Jun 15;245(1-2):67-72. doi: 10.1016/j.jns.2005.05.020. Epub 2006 Apr 19. PMID 16626751
- [Background] Benedict RH, Ramasamy D, Munschauer F, Weinstock-Guttman B, Zivadinov R. Memory impairment in multiple sclerosis: correlation with deep grey matter and mesial temporal atrophy. J Neurol Neurosurg Psychiatry. 2009 Feb;80(2):201-6. doi: 10.1136/jnnp.2008.148403. Epub 2008 Oct 1. PMID 18829629
- [Background] Foong J, Rozewicz L, Quaghebeur G, Thompson AJ, Miller DH, Ron MA. Neuropsychological deficits in multiple sclerosis after acute relapse. J Neurol Neurosurg Psychiatry. 1998 Apr;64(4):529-32. doi: 10.1136/jnnp.64.4.529. PMID 9576548
- [Background] Feuillet L, Reuter F, Audoin B, Malikova I, Barrau K, Cherif AA, Pelletier J. Early cognitive impairment in patients with clinically isolated syndrome suggestive of multiple sclerosis. Mult Scler. 2007 Jan;13(1):124-7. doi: 10.1177/1352458506071196. PMID 17294621
- [Background] Glanz BI, Holland CM, Gauthier SA, Amunwa EL, Liptak Z, Houtchens MK, Sperling RA, Khoury SJ, Guttmann CR, Weiner HL. Cognitive dysfunction in patients with clinically isolated syndromes or newly diagnosed multiple sclerosis. Mult Scler. 2007 Sep;13(8):1004-10. doi: 10.1177/1352458507077943. Epub 2007 Jul 10. PMID 17623735
- [Background] Simmons RD, Tribe KL, McDonald EA. Living with multiple sclerosis: longitudinal changes in employment and the importance of symptom management. J Neurol. 2010 Jun;257(6):926-36. doi: 10.1007/s00415-009-5441-7. Epub 2010 Jan 19. PMID 20084515
- [Background] Benedict RH, Zivadinov R. Risk factors for and management of cognitive dysfunction in multiple sclerosis. Nat Rev Neurol. 2011 May 10;7(6):332-42. doi: 10.1038/nrneurol.2011.61. PMID 21556031
- [Background] Patti F, Pozzilli C, Montanari E, Pappalardo A, Piazza L, Levi A, Onesti E, Pesci I; Italian Study Group On Quality Of Life In Ms. Effects of education level and employment status on HRQoL in early relapsing-remitting multiple sclerosis. Mult Scler. 2007 Jul;13(6):783-91. doi: 10.1177/1352458506073511. Epub 2007 Feb 16. PMID 17613607
- [Background] Amato MP, Ponziani G, Rossi F, Liedl CL, Stefanile C, Rossi L. Quality of life in multiple sclerosis: the impact of depression, fatigue and disability. Mult Scler. 2001 Oct;7(5):340-4. doi: 10.1177/135245850100700511. PMID 11724451
- [Background] Amato MP, Ponziani G, Siracusa G, Sorbi S. Cognitive dysfunction in early-onset multiple sclerosis: a reappraisal after 10 years. Arch Neurol. 2001 Oct;58(10):1602-6. doi: 10.1001/archneur.58.10.1602. PMID 11594918
- [Background] Morrow SA, Jurgensen S, Forrestal F, Munchauer FE, Benedict RH. Effects of acute relapses on neuropsychological status in multiple sclerosis patients. J Neurol. 2011 Sep;258(9):1603-8. doi: 10.1007/s00415-011-5975-3. Epub 2011 Mar 8. PMID 21384163
- [Background] Benedict RH, Fischer JS, Archibald CJ, Arnett PA, Beatty WW, Bobholz J, Chelune GJ, Fisk JD, Langdon DW, Caruso L, Foley F, LaRocca NG, Vowels L, Weinstein A, DeLuca J, Rao SM, Munschauer F. Minimal neuropsychological assessment of MS patients: a consensus approach. Clin Neuropsychol. 2002 Aug;16(3):381-97. doi: 10.1076/clin.16.3.381.13859. PMID 12607150
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] Smith A. Symbol digit modalities test: Manual. Los Angeles: Western Psychological Services, 1982.
- [Background] Benedict R. Brief Visuospatial Memory Test - Revised: Professional Manual. Odessa, Florida: Psychological Assessment Resources, 1997.
- [Background] Gronwall DM. Paced auditory serial-addition task: a measure of recovery from concussion. Percept Mot Skills. 1977 Apr;44(2):367-73. doi: 10.2466/pms.1977.44.2.367. PMID 866038
- [Background] Benedict RH, Bruce J, Dwyer MG, Weinstock-Guttman B, Tjoa C, Tavazzi E, Munschauer FE, Zivadinov R. Diffusion-weighted imaging predicts cognitive impairment in multiple sclerosis. Mult Scler. 2007 Jul;13(6):722-30. doi: 10.1177/1352458507075592. Epub 2007 Mar 15. PMID 17613599
- [Background] Benedict RH, Holtzer R, Motl RW, Foley FW, Kaur S, Hojnacki D, Weinstock-Guttman B. Upper and lower extremity motor function and cognitive impairment in multiple sclerosis. J Int Neuropsychol Soc. 2011 Jul;17(4):643-53. doi: 10.1017/S1355617711000403. PMID 21486517
- [Background] Filippini G, Brusaferri F, Sibley WA, Citterio A, Ciucci G, Midgard R, Candelise L. Corticosteroids or ACTH for acute exacerbations in multiple sclerosis. Cochrane Database Syst Rev. 2000;2000(4):CD001331. doi: 10.1002/14651858.CD001331. PMID 11034713
- [Background] Shah A, Eggenberger E, Zivadinov R, Stuve O, Frohman EM. Corticosteroids for multiple sclerosis: II. Application for disease-modifying effects. Neurotherapeutics. 2007 Oct;4(4):627-32. doi: 10.1016/j.nurt.2007.07.009. PMID 17920543
- [Background] Frohman EM, Shah A, Eggenberger E, Metz L, Zivadinov R, Stuve O. Corticosteroids for multiple sclerosis: I. Application for treating exacerbations. Neurotherapeutics. 2007 Oct;4(4):618-26. doi: 10.1016/j.nurt.2007.07.008. PMID 17920542
- [Background] Fischer JS, Rudick RA, Cutter GR, Reingold SC. The Multiple Sclerosis Functional Composite Measure (MSFC): an integrated approach to MS clinical outcome assessment. National MS Society Clinical Outcomes Assessment Task Force. Mult Scler. 1999 Aug;5(4):244-50. doi: 10.1177/135245859900500409. PMID 10467383
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Benedict RHB, Schretlen D, Groninger L, Dobraski M, Shpritz B. Revision of the Brief Visuospatial Memory Test: Studies of normal performance, reliability, and validity. Psychological Assessment 8:145-153, 1996.
- [Background] Benedict RH, Munschauer F, Linn R, Miller C, Murphy E, Foley F, Jacobs L. Screening for multiple sclerosis cognitive impairment using a self-administered 15-item questionnaire. Mult Scler. 2003 Feb;9(1):95-101. doi: 10.1191/1352458503ms861oa. PMID 12617275
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Gilson BS, Gilson JS, Bergner M, Bobbit RA, Kressel S, Pollard WE, Vesselago M. The sickness impact profile. Development of an outcome measure of health care. Am J Public Health. 1975 Dec;65(12):1304-10. doi: 10.2105/ajph.65.12.1304. No abstract available. PMID 1200192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Started | 30 | 34
Completed | 29 | 32
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: The sample used for final analysis was smaller than the total enrolled (see Participant Flow) because participants were excluded from the final analysis due to (1) withdrawal prior to follow-up, (2) occasional missing data from one or more timepoints, and (3) to optimize matching of the groups based on demographic characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (10.7) | 43.8 (10.5) | 43.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Symbol Digit Modalities Test [Mean (Standard Deviation); unit: Total Correct] — A measure of visual processing speed and working memory. Minimum score of 0, Maximum score of 120. Higher scores indicate better performance.
  Total Correct | 55.2 (13.5) | 55.9 (12.4) | 55.6 (13.0)
California Verbal Learning Test, 2nd Edition [Mean (Standard Deviation); unit: Total Learning Score] — Measure of verbal memory. Minimum 0, Maximum 60. Higher scores indicate better performance.
  Total Learning Score | 51.4 (12.6) | 49.1 (11.1) | 50.3 (11.9)
Brief Visuospatial Memory Test Revised (BVMTR) [Mean (Standard Deviation); unit: Total Learning Score] — A measure of visual-spatial memory. Minimum of 0, maximum of 36. Higher scores indicate better performance.
  Total Learning Score | 23.1 (7.1) | 23.9 (7.0) | 23.5 (7.1)
Timed 25-foot Walk [Mean (Standard Deviation); unit: Seconds] — Measure of walking speed and ambulation, how fast can a subject walk 25 feet, measured in seconds. Ceiling value of 300 seconds.
  Seconds | 5.4 (1.9) | 5.0 (1.2) | 5.2 (1.6)
Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ) [Mean (Standard Deviation); unit: Total Score] — Self-report measure of neuropsychological impairment. Minimum of 0, maximum of 60. Higher scores indicate greater self-reported neuropsychological impairment.
  Total Score | 30.1 (12.6) | 18.0 (8.9) | 24.1 (10.8)
Expanded Disability Status Scale (EDSS) [Median (Inter-Quartile Range); unit: Total Score] — A clinician assigned measure of disability specific to MS. Minimum of 0 (no disability), maximum of 10 (death due to MS). Higher scores indicate greater disability.
  Total Score | 2.5 [2.0 to 3.5] | 2.5 [1.75 to 3.0] | 2.5 [1.75 to 3.5]
Fatigue Severity Scale (FSS) [Mean (Standard Deviation); unit: Total Score] — Self-report measure of fatigue on 1 (minimum) to 9 (severe fatigue) scale.
  Total Score | 4.9 (1.6) | 4.2 (1.5) | 4.6 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Symbol Digit Modalities Test (SDMT)
Description: A measure of visual processing speed and working memory. Minimum score of 0, Maximum score of 120. Higher scores indicate better performance. The difference in total correct responses on the SDMT from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Correct
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Correct | 44.6 (13.9) | 58.5 (13.9)

2. Primary Outcome: Timed 25-foot Walk
Description: An MS-specific measure of functional status walking speed. How many seconds does it take to walk 25 feet. Ceiling value of 300 seconds.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Seconds | 6.7 (3.2) | 5.3 (1.2)

3. Primary Outcome: Change From Baseline on the Paced Auditory Serial Addition Test (PASAT)
Description: A measure of auditory processing speed and working memory. Minimum value of 0, maximum value of 60. Higher score indicates better performance. The difference in total correct on the PASAT from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Correct
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Correct | 40.1 (12.2) | 47.0 (14.3)

4. Primary Outcome: Change From Baseline on the Brief Visuospatial Memory Test-Revised (BVMT-R)
Description: A measure of visual/spatial memory. Minimum of 0, maximum of 36. Higher score indicates better performance. The difference in total learning score on the BVMT-R from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Learning Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Learning Score | 22.0 (8.9) | 22.5 (7.9)

5. Primary Outcome: Change From Baseline on the California Verbal Learning Test, Second Edition (CVLT-II)
Description: A measure of auditory/verbal episodic memory. Minimum of 0, maximum of 80. Higher score indicates better performance. The difference in total learning score on the CVLT-II from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Learning Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Learning Score | 46.6 (14.1) | 51.2 (11.8)

6. Secondary Outcome: Change From Baseline on the Expanded Disability Status Scale (EDSS).
Description: A clinician assigned measure of disability specific to MS. Minimum of 0 (no disability), maximum of 10 (death due to MS). Higher scores indicate greater disability. The difference in total score on the EDSS from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Total Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Score | 3.0 [2.0 to 3.5] | 2.0 [1.5 to 3.25]

7. Secondary Outcome: Change From Baseline on the Multiple Sclerosis Neuropsychological Questionnaire (MSNQ)
Description: A self and informant rating measure of perceived cognitive problems. Minimum of 0, maximum of 60. Higher scores indicates greater self-reported neuropsychological impairment. The difference in total score on the MSNQ from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Score | 34.5 (9.4) | 20.0 (12.3)

8. Secondary Outcome: Change From Baseline on the Beck Depression Inventory-Fast Screen (BDI-FS)
Description: A self-report, multiple choice inventory of depression. Minimum of 0, maximum of 21. Higher score indicates higher levels of depression. The difference in total score on the BDI-FS from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Score | 5.0 (4.0) | 1.6 (2.8)

9. Secondary Outcome: Change From Baseline on the Fatigue Severity Scale (FSS)
Description: A self-report measure of fatigue. 1 (no fatigue) to 9 (severe fatigue). The difference in total score on FSS from Day 0 to Day 90 were analyzed to address change in this outcome.
Time Frame: Day 0 and Day 90
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
Number analyzed (Participants) | 25 | 25
Total Score | 5.4 (1.4) | 3.8 (1.7)

10. Other Pre Specified Outcome: Incidence of Adverse Events
Description: The number of patients reporting adverse events over the course of the study
Time Frame: Up to 3 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change From Baseline in Concurrent Medications
Description: Initiation or discontinuation of any medications occurring over the course of the study; monitored by clinician and study personnel.
Time Frame: Up to 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For individual subjects the time period was 3 months. From the initial enrollment to study closure, total monitoring time was 4 years.
Description: At each visit and in the weeks between visits, subjects were asked if they were experiencing any adverse events.
Arm/Group | Cognitively Relapsing Patients | Stable Multiple Sclerosis Patients
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Because of withdrawals and/or incomplete data, some enrolled subjects were excluded from the final data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT02290444/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT02290444/ICF_001.pdf